CLINICAL TRIAL: NCT03191214
Title: An Observational Thermography Study of the Core-peripheral Temperature Gradient as a Function of Vascular Resistance During the Redistribution Phase Following the Induction of General Anaesthesia in Warmed and Non-warmed Patients
Brief Title: Impact of Forced Air Warming on Perioperative Thermodynamics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 228666
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Hypothermia Following Anesthesia
Keywords: Infra-red thermography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- No Warming: Patients undergoing brief surgical procedures of >15 minutes for whom no warming devices are being employed.
- Forced Air Warming: Patients undergoing surgical procedures in which forced air warming, is being used
  Interventions: Device: Intraoperative Forced Air Warming

INTERVENTIONS:
Device: Intraoperative Forced Air Warming — As part of their standard care, patients undergoing surgery >30 min in duration will receive forced air warming in the form of a Bair Hugger. This is a blanket covering their upper torso and arms into which warm air is blown.
  Groups: Forced Air Warming

SUMMARY:
The purpose of the study is to assess the temperature changes that take place throughout the body in a real world setting, when a patient is given general anaesthesia. Specifically we will investigate the movement of body heat from the core to the peripheries at the beginning of surgery. This will be measures with a series of temperature sensors and infrared thermography

DETAILED DESCRIPTION:
Intra-operative hypothermia increases the risk of a wide range of post operative complications; wound infection, damage to heart muscle, and an increased length of hospital stay.

A range of technologies exist for maintaining the temperature of patients undergoing surgical procedures. Yet despite the frequent use of forced air warming devices, a significant reduction in core temperature can occur in the first 60 minutes of some major surgeries.

This is an Observational Cross-Sectional Study, investigating patients undergoing elective surgery in two groups Group 1: Patients undergoing brief surgical procedures of >15 minutes for whom no warming devices are being employed.

Group 2: Patients undergoing surgical procedures in which forced air warming, is being used Potential participants will first be approached by medical staff at their pre-operative assessment clinic. They will be screened for exclusion criteria before being given a participant information sheet, which will be explained to them. They will be invited to contact the researcher if they are interested in participating in the study.

On arrival in hospital the day of their surgery, the patients will be met by their anaesthetist and a researcher who will provide any further information required about the study, and consent will be taken.

Following receipt of informed consent, patients will be involved from 30 minutes before their surgery begins, until the end of their surgery.

The null hypothesis is that there is no difference in the rate of flow of heat from the core to the peripheries between patients who receive warming during surgery, and those who do not. As it would be unethical to randomise a patient to not receive warming, we have designed an observational study to compare patients who are warmed / not warmed as part of their standard care. Patients undergoing surgery <30 minutes long are not routinely warmed during surgery.

Potential participants will be informed of the study at the pre-operative assessment clinic in the weeks preceding surgery. Posters will be located in the clinic rooms and relevant areas, and subjects will be given information by the clinic staff to read prior to their surgery.

Participants will be admitted to hospital the evening prior, or the morning of surgery, whereupon they will undergo standard admission processes, including pre-operative assessment by the anaesthetist assigned to that list. The anaesthetist and researcher will then explain the study again, reiterating the potential risks and benefits of the study to the patient themselves, and to the population as a whole. Written consent will be sought at this point.

Participants will be weighed and four measurements will be taken, comprising : arm length, leg length, trunk length and maximum abdominal width. Participants will stand onto a bioimpedance machine, which will quantify their body fat and body water percentage.

30 minutes before their operation, skin temperature sensors will be placed on the patient's forehead, forearm, finger, hip, calf and toe. An additional SpotOn temperature sensor, placed on the forehead will be used to non invasively measure core temperature.

Measurement of blood pressure, cardiac output and systemic vascular resistance will be obtained by a finger cuff connected to a Nexin Noninvasive cardiac output monitor. These measurements describe the action of the heart and blood vessels. At the end of each surgery the data recorded on this device will be transferred via an encrypted USB key onto a data acquisition laptop.

Temperature measurements from the seven of sensors will taken at 5 second intervals onto a data acquisition laptop.

At 15 minutes intervals Infra red thermography images will be taken from a FLIR a320 device. This equipment will be mounted on a raised boom above the surgeons, in a sterile sleeve. This will not be held over the patient at any point, and will be moved away from the patient between measurements.

Once the surgery has ended, and the patient has been transferred to the recovery area, all temperature sensors will be removed and the patient will exit the trial.

A sample size of 24 patients will be recruited to quantify the effect of warming.

ELIGIBILITY:
Inclusion Criteria:

* Male & Female patients, from 18 - 80 years old, undergoing surgery requiring general anaesthesia, who are deemed to have capacity to give informed consent and have done so in writing prior to commencement of surgery.

The surgeries include :

1. brief surgical procedures of >15 minutes requiring general for whom no warming devices are being employed
2. surgical >30 minutes procedures in which forced air warming, is being used

Exclusion Criteria:

Patients who do not adequately understand verbal explanations or written information given in English.

Patients not possessive of capacity to give informed consent. Patients who have not given consent.

Patients with :

* Peripheral vascular disease
* BMI >30
* Aortic aneurysms
* Amputations

Patients with a history of:

* Thyroid disease
* Dysautonomia
* Malignant hyperthermia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2017-07-21 (Estimated); Primary Completion 2017-09-15 (Estimated); Study Completion 2017-09-15 (Estimated)

PRIMARY OUTCOMES:
The change in core - peripheral temperature gradient | At 25 minutes following induction of anaesthesia
  This will be calculated as the sum of, the increase in peripheral temperature and the decrease in core temperature, between 0 and 25 minutes from the induction of anaesthesia.
  Peripheral temperature will be determined by segmental thermal analysis of thermography data, calibrated against skin temperature sensors.

SECONDARY OUTCOMES:
Peripheral to core heat transfer due to warming | Between 60 minutes and 120 minutes following induction of anaesthesia
  The increase in core temperature at 120 minutes compared to 60 minutes, as a proportion of the increase in temperature induced in the peripheries being warmed, over the same time period.
Change in temperature gradient as a function of time & systemic vascular resistance | For the first 25 minutes following induction of anaesthesia
  Changes in the core peripheral temperature gradient (detailed in the 1º outcome) will be fitted as a function of time and systemic vascular resistance. The coefficients of this function will be compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Fintan Hughes, Study Director — Univeristy College London Hospital
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No